CLINICAL TRIAL: NCT00651729
Title: Safety Study of Botulinum Toxin Type A for the Treatment of Focal Upper Limb Poststroke Spasticity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191622-056
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Stroke; Muscle Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A

ARMS (1):
- 1 (Experimental): Botulinum Toxin Type A
  Interventions: Biological: Botulinum Toxin Type A

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Each patient received from 1 to 5 treatments, with a minimum of 12 weeks between treatments. For each treatment, a total dose of 200 U to 400 U botulinum toxin Type A was injected into the wrist and finger flexor muscles of the affected upper limb, not to exceed 6 U/kg
  Other Names: BOTOX®

SUMMARY:
The purpose of this study is to evaluate the safety of repeated doses of Botulinum Toxin Type A for the treatment of focal upper limb poststroke spasticity

ELIGIBILITY:
Inclusion Criteria:

* Medically stable poststroke patients with spastic muscles in the upper limb

Exclusion Criteria:

* Stroke within 6 months of study enrollment
* Previous therapy with Botulinum Toxin Type A for treatment of any condition prior to 4 months of enrollment, for treatment of any condition prior to 01 January 1998

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2003-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | Week 54

SECONDARY OUTCOMES:
Spasticity as measured by the Ashworth scale | Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Indianapolis, Indiana, United States
- Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Elovic EP, Barron RL, Liu J, Turkel CC. Resource utilization, productivity, and caregiver burden impact in a trial of repeated doses of botulinum toxin type A for the treatment of focal upper-limb poststroke spasticity: A multicenter open-label study. Arch Phys Med Rehabil 2005;86(9):E46 ABS-Poster 239
- [Background] Elovic EP, Brashear A, Kaelin D, McIntosh R, Liu J, Turkel CC. Safety and efficacy of repeated botulinum toxin type A treatments for focal upper-limb poststroke spasticity: Results of a 12-month multicenter, open-label trial. Arch Phys Med Rehabil 2005,86(9):E46-7 ABS-Poster 242.
- [Background] Mayer N, Barron RL, Liu J, Turkel CC. The burden of illness associated with loss of function after stroke in patients with arm spasticity enrolled in a multicenter open-label study. Arch Phys Med Rehabil 2005;86(9):E47 ABS-Poster 243
- [Background] Childers MK, Barron RL, Patel RK, Turkel CC. Health utility and quality of life following botulinum toxin type A in repeated doses for the treatment of focal upper-limb spasticity in stroke patients: A multicenter open-label study. Arch Phys Med Rehabil 2005;86(9):E48 ABS-Poster 249
- [Background] Mayer N, Barron R, Liu J, Turkel C. The burden of illness associated with loss of function after stroke in patients with arm spasticity enrolled in a multicenter open-label study. Arch Phys Med Rehabil 2006 Oct;87(10):E46-7 POS-Poster 54.
- [Background] Elovic E, Kaelin D, Brashear A, McIntosh R, Liu J, Barron R. Safety and efficacy of repeated botulinum toxin type A for focal upper-limb poststroke spasticity in patients aged 65 and older in a 12-month multicenter open-label trial. Arch Phys Med Rehabil 2006 Oct;87(11):E50 ABS-PR_272
- [Background] Elovic E, rashear A, Kaelin D, Abu-shakra S, VanDenburgh A, Turkel CC, Beddingfield III F. The effect of repeated treatment of botulinum toxin type A on poststroke, spasticity-related pain: A subgroup analysis of patients in a 12-month trial. Arch Phys Med Rehabil 2007 Sep;88(10):E4 ABS-Article 13.
- [Background] Elovic E, Brashear A, Kaelin D, Liu J, VanDenburgh AM, Beddingfield III F. The effect of repeated treatment of botulinum toxin type A on poststroke, spasticity-related pain: A subgroup analysis of patients in a 12-month trial. Arch Phys Med Rehabil 2007 Sep;88(9):E65 ABS-Poster 195
- [Background] Childers MK, Barron RL, Patel RK, Turkel CC. A multi-center open label study of botulinum toxin type A (BoNT/A) treatment of focal upper limb post-stroke spasticity: Health utility and quality of life assessment. Can Assoc Phys Med & Rehabil Annual Meeting 2006;(Online):ABS-CL-47
- [Background] Elovic E, Barron RL, Lui J, Turkel CC. Repeated doses of botulinum toxin type A (BoNT/A) for the treatment of post-stroke focal upper limb spasticity: Assessments of resource utilization, caregiver burden, and productivity. Can Assoc Phys Med & Rehabil Annual Meeting 2006;(Online):ABS-CL-49
- [Background] Elovic E, Brashear A, Kaelin D, McIntosh R, Lui J, Turkel C. Assessment of safety and efficacy of multiple botulinum toxin type A (BoTN/A) injections for post-stroke focal upper limb spasticity: A one year-long multicenter, open-label trial. Can Assoc Phys Med & Rehabil Annual Meeting 2006;(Online):ABS-CL-51
- [Background] Elovic E, Brashear A, Kaelin D, McIntosh R, Liu J, Turkel CC. Safety and efficacy of repeated botulinum toxin type A (BoNTA) in the treatment of poststroke, upper limb spasticity: A 12-month trial. Mov Disord 2006;21(Suppl 15):S423 ABS-P347
- [Background] Elovic E, Brashear A, Kaelin D, McIntosh R, Liu JY, Barron R, Turkel C. Safety and efficacy of repeated botulinum toxin type A for focal upper limb poststroke spasticity in patients aged 65 years and older in a 12-month multicenter open-label trial. Neurology 2006 14 Mar;66(5 Suppl 2):A297-8 ABS-P05.156
- [Background] Slavic E, Brashear A, Kaelin D, McIntosh R, Liu J, Turkel C. The effect of repeated treatment of botulinum toxin type A on poststroke, spasticity-related pain: A subgroup analysis of patients in a 12-month trial. Neurology 2007;68(12 Suppl 1):A177 ABS-P04.131
- [Background] Elovic E, Brashear A, Kaelin D, McIntosh R, Liu J, Turkel C. Safety and efficacy of repeated botulinum toxin type A treatments for focal upper limb poststroke spasticity: Results of a 12-month multicenter, open-label trial. Neurotox Res 2006 Apr;9(2-3):230 ABS-P23
- See also: Link to Clinical Trial Results — http://www.allerganclinicaltrials.com